CLINICAL TRIAL: NCT04502108
Title: Online Survey About Physical Activity and Nutrition During and After Coronavirus Pandemic
Brief Title: Behavior During and After COVID-19 Crisis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Slavko Rogan (Other)
Responsible Party: Sponsor-Investigator, Slavko Rogan, University lecturer, Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Other Study IDs: BFH Corona
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Exercise; Nutritional Status; Sleep
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Employees: Employees of the Department of Health Professions, Bern University of Applied Sciences
  Interventions: Behavioral: Covid19
- Students: Students of the Department of Health Professions, Bern University of Applied Sciences
  Interventions: Behavioral: Covid19

INTERVENTIONS:
Behavioral: Covid19 — Impact of the COVID19-pandemic on physical activity, nutritional habits and sleeping behavior during an extraordinary period of confinement and social distancing, during the loosening phase and social distancing and the phase after the pandemic.

SUMMARY:
A crisis situation leads to changes in life. During December 2019, many people contracted pneumonia in the Chinese city of Wuhan. On January 7, 2020, the novel coronavirus (Covid-19) was identified as the cause of this disease. Within five months, the virus spread around the globe and forced countries to restrict public life. Due to the high infection rates in Europe, a lockdown followed between March and April 2020 (except in Sweden). As the number of infections decreased, European countries began to gradually relax the lockdown from May 2020.

The lockdown and the later stages of loosening have an impact on lifestyle. Institutions of higher education must also adapt to this situation and have switched to distance learning.

The University of Applied Sciences of Bern (BFH), Department of Health Professions with the Departments (DHP) of Nutrition and Dietetics and Physiotherapy, considers the question of the degree to which nutritional and exercise behavior has changed.

The findings provide recommendations for future crises for students and employees of the BFH-DHP.

In order to achieve this, at the BFH-DHP two anonymous online surveys will be conducted.

DETAILED DESCRIPTION:
There is little evidence of how physical activity and eating behavior changes during a pandemic period and in the period after a pandemic period of students and employees at the BFH-DHP. This observational study will assists to determine the impact of an immediate change within a pandemic on physical activity, nutrition, sleep and alcohol consumption and the consequences after a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Students from the Bern University of Applied Sciences, Department of Health Professions
* Students from the Bern University of Applied Sciences, Department of Health Professions

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All students and employees from the Bern University of Applied Sciences, Department of Health Professions participating in the study will be invited to answer the online survey. The sample will include students in different academic degrees: bachelor's degree and master's degree and from different study degree courses (midwife, nurse, nutrition and dietetics and physiotherapy) and employees.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity 2020 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period
  Mean number of minutes spent physically active (standing, walking, running) per day. A validated German short version of the international physical activity questionnaire (iPAQ-SF) will be used to assess physical activity over the last seven days
Physical activity 2021 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period in 2021
  Mean number of minutes spent physically active (standing, walking, running) per day. A validated German short version of the international physical activity questionnaire (iPAQ-SF) will be used to assess physical activity over the last seven days

SECONDARY OUTCOMES:
Nutrition 2020 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period
  Mean number of habitual food and nutrient intake per day
Nutrition 2021 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period in 2021
  Mean number of habitual food and nutrient intake per day
Alcohol 2020 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period
  Liters of pure alcohol per day
Alcohol 2021 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period in 2021
  Liters of pure alcohol per day
Sleep 2020 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period
  Average number of hours of sleep during the night
Sleep 2021 | During COVID-19 pandemic crisis: the survey will be conducted within an one month period in 2021
  Average number of hours of sleep during the night

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Baur, Ph.D, Principal Investigator — BFH, Department of Health Professions, Faculty of Physiotherapy
Locations (1):
- Bern University of Applied Sciences, Department of Health Professions, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Due to the anonymous data collection, there will be no individual participants' data available. The study protocol will be published in an internationally recognized journal.

REFERENCES:
- [Derived] Taeymans J, Luijckx E, Rogan S, Haas K, Baur H. Physical Activity, Nutritional Habits, and Sleeping Behavior in Students and Employees of a Swiss University During the COVID-19 Lockdown Period: Questionnaire Survey Study. JMIR Public Health Surveill. 2021 Apr 13;7(4):e26330. doi: 10.2196/26330. PMID 33630747
- [Derived] Rogan S, Luijckx E, Taeymans J, Haas K, Baur H. Physical Activity, Nutritional Habits, and Sleep Behavior Among Health Profession Students and Employees of a Swiss University During and After COVID-19 Confinement: Protocol for a Longitudinal Observational Study. JMIR Res Protoc. 2020 Dec 22;9(12):e25051. doi: 10.2196/25051. PMID 33296868